CLINICAL TRIAL: NCT03749135
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Proof-of-concept Phase 2, 16-week Treatment Study With a 16 Week Follow-up Period to Assess the Efficacy and Safety of Dupilumab (Anti-IL4Ra) in Adult Patients With Chronic Spontaneous Urticaria Despite H1-antihistamine Treatment.
Brief Title: Dupilumab in Chronic Spontaneous Urticaria
Acronym: DUPICSU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Sanofi (Industry); Proinnovera GmbH (Industry)
Responsible Party: Principal Investigator, Marcus Maurer, Research Director Prof. Dr. med. Marcus Maurer, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-001-01; 2017-004458-41 (EudraCT Number)
Record Dates: First submitted 2018-07-12; First posted 2018-11-21 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Chronic Spontaneous Urticaria; Recurrent Angioedema
Keywords: hives; itch
MeSH Terms: conditions — Chronic Urticaria; Angioedema; Urticaria; Pruritus | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: This is a Phase 2a multicenter, randomized, double blind, placebo controlled, parallel group, two-arm, proof-of-concept investigator-initiated trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupilumab (Active Comparator): Dupilumab (anti-IL4Ra), s.c. administration
  Interventions: Drug: Dupilumab
- Placebo Comparator (Placebo Comparator): matching Placebo, s.c. administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — anti-IL4-Receptor alpha
  Arms: Dupilumab
Drug: Placebo — Placebo
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to assess the efficacy in reducing disease activity and safety of Dupilumab in adult patients with chronic spontaneous urticaria (CSU) who are symptomatic despite H1-antihistamine treatment.

DETAILED DESCRIPTION:
Treatment with Dupilumab has been shown to reduce clinically significant exacerbations and to improve skin symptom control as well as quality of life in moderate to severe atopic dermatitis patients and in moderate to severe asthma patients. It has been approval by European Medicines Agency (EMA) for the treatment of atopic dermatitis patients in September 2017.

Dupilumab is a novel monoclonal antibody that inhibits interleukin-4 (IL-4) and interleukin-13 (IL-13) signaling and was previously found to be effective in atopic dermatitis and asthma. Considering that CSU and atopic diseases share many common features (e.g. key pathogenic role of mast cells and immunoglobulin E (IgE), itch is a dominant symptom, Th2 dominance), it is reasonable to expect that Dupilumab is beneficial in CSU.

These results suggest that Dupilumab may provide an effective treatment option for patients with insufficient treatment responses to H1-antihistamines exhibiting wheal and flare type skin reactions.

The gold standard treatment of CSU consists of administration of antihistamines. In more than 50% of the patients, symptoms persist with standard dosing of antihistamines. In antihistamine-refractory patients with chronic spontaneous urticaria, the currently only licensed treatment is omalizumab, a monoclonal anti-IgE antibody. In 2014, omalizumab has been licensed for add-on therapy in CSU patients who still have symptoms despite standard-dosed antihistamine treatment. There is, however, still a great medical need for additional treatment options, as 20-40% of patients are still without effective therapy. These patients have no other licensed treatment option and can only be treated off-label with therapeutics with several known safety risks such as Cyclosporine A.

Dupilumab has excellent potential to provide symptom control in CSU. This study will provide additional valuable insights into the therapeutic potential of Dupilumab in improving quality of life in these patients, in addition to managing CSU symptoms.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis: chronic spontaneous urticaria (defined as ongoing disease)

1. Patient is informed about study procedures and medications and has given written informed consent before any assessment.
2. Patient is able to communicate with the investigator, understands and complies with the requirements of the study.
3. Male or Female
4. Patient is 18-75 years of age
5. Patient is diagnosed with moderate to severe CSU and refractory to standard of care treatment at the time of randomization, as defined by the following:

   1. The presence of itch and hives for more than 6 consecutive weeks at any time prior to enrollment despite current use of H1 antihistamine
   2. Urticaria activity score UAS7 score (range 0-42) equal or more than 16, 7 days prior to randomization (Day 1)
   3. CSU diagnosis for 6 months
6. Willing and able to complete a daily symptom diary for the duration of the study and adhere to the study visit schedules.
7. Patients must not have more than one missing diary entry in the 7 days prior to randomization. Re-screening may be considered.
8. Women of childbearing potential have to agree to use an acceptable form of contraception (as determined by the site investigator) and have to continue its use for the duration of the study.

Exclusion Criteria:

1. Patients whose urticaria is solely due to inducible urticaria.
2. Other diseases with symptoms of urticaria or angioedema, including urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa), and hereditary or acquired angioedema (e.g., due to C1 inhibitor deficiency)
3. Any other active skin disease associated with chronic itching that might confound the study evaluations and results (e.g., atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, etc.)
4. Patients who have received concomitant prohibited medication within the last 3 months prior to screening

   * Anti-IgE therapy (e.g. omalizumab)
   * Routine (daily or every other day during 5 or more consecutive days) doses of systemic corticosteroids or other immunosuppressants
   * Intravenous immunoglobulins
   * Biological therapy
   * Systemic immunosuppressants
   * Live/attenuated vaccines
   * Other investigational drug
5. History of anaphylactic shock
6. Active helminthic parasite infection or treatment of helminthic parasites within 6 months of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Urticaria activity score over 7 days (UAS7) | Change from 7 days prior to baseline (Visit (V) 1) to 7 days prior to week 16 (V9)
  0-42 Points total range over 7 days, higher values equal more disease activity

SECONDARY OUTCOMES:
Itch severity score (ISS7; 0 - no pruritus; 21 - most severe pruritus), hive severity score (HSS7; 0 - no hives; 21 - max. hive severity) | Change from 7 days prior to baseline (Visit (V) 1) to 7 days prior to week 16 (V9)
  Disease activity scores
Global assessment for disease activity | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)
  Global assessment for disease activity(physician and patient) by visual analogue scale (VAS; 0 - no pain; 10 - max. amount of pain)
urticaria control test (UCT; 16 - complete disease control; 0 - strong symptoms), dermatological quality of life (DLQI; 0 - no impairment; 30 - max. impairment), chronic urticaria quality of life (Cu2-QoL; 23 - no impairment; 115 - max. impairment) | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)
  Disease specific quality of life
Responder rates (regarding disease activity and quality of live (QoL)) | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)
  Responder rates (regarding disease activity and quality of live (QoL))
rate of angioedema burdened days angioedema activity score (AAS; 0 - lowest disease activity; 15 - highest disease activity) angioedema quality of life (AE-Qol; 0 - no impairment; 100 - worst impairment) | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)]
  For patients with concomitant angioedema
Rescue medication use | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)]
  Frequency of of how often rescue medication is used

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (6):
- Germany (6):
  - Universitätsklinikum Giessen und Marburg, Marburg, Hesse
  - Hautklinik Universitätsklinikum Münster, Münster, NRW, Germany
  - Hautklinik der Universitätsmedizin Mainz Clinical Research Center, Mainz, Rheinland-Pfalz, Germany
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsmedizin Leipzig, Klinik für Dermatologie, Venerologie und Allergologie, Leipzig, Saxony
  - Charite University, Berlin, Germany, Berlin

IPD SHARING:
Plan to Share IPD: No